CLINICAL TRIAL: NCT05884788
Title: Study of the Life Stories of Patients Making a Request for Euthanasia, in the Context of Advanced Cancer.
Acronym: RECIFE
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET22000324
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer
Keywords: Euthanasia; Cancer
MeSH Terms: conditions — Suicide, Assisted; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: free interview, and questionnaires in a second time — After inclusion in the study, patients will be met for a free interview. The interview will be conducted using an open-ended interview method with the patients to allow free expression of their life history, using open and broad questions to avoid the influence of the interviewer as much as possible.
  Each interview will be conducted by the same person to allow for better interpersonal reproducibility.
  After the interview, the patients will be seen again to complete two questionnaires:
  * An attachment questionnaire: Relationship Scales Questionnaire
  * A questionnaire on symptoms: Distress thermometer

SUMMARY:
This study wishes to focus on the life course of patients, beyond the moments of suffering experienced at the time of the request for euthanasia. It is based on the perspective that the patient's account of his or her life course can be a source of information for better understanding and accompanying patients requesting euthanasia.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* With cancer in the palliative phase, i.e. with an incurable disease according to current knowledge.
* Expressing a request for euthanasia in terms evoking a request for death with the intervention of an outside person.
* Non-opposition to the study after full written information.

Exclusion Criteria:

* Severe decompensated psychiatric pathology
* Vulnerable persons defined here as pregnant women, parturients and persons under legal protection or unable to express their consent
* Inability to conduct an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conduct our study in a French cancer center and a French public hospital. Patients requesting euthanasia will be informed about the possibility of participating in our study. If the patients agree, and if they meet the study criteria, they will be included.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Description of the life stories of patients requesting euthanasia to explore which life experiences are brought forward when making this request, in a context of advanced oncological pathology. | One month
  The main objective is to describe the life stories of patients requesting euthanasia in order to discover which life experiences are reasoning in the formulation of this request, in a context of advanced oncological pathology.
  The investigators carry out a descriptive analysis of the interviews. The interviews will be analyzed as they are conducted, in order to identify themes of interest. The themes will be compared between the different interviews in order to identify possible trends.

SECONDARY OUTCOMES:
Calculation of the Bartholomew score | One month
  Use of specific questionnaire (Relationship Scales Questionnaire of Batholomew) to describe the profiles of the patients in the study
Calculation of the distress thermometer's score | One month
  Use of specific questionnaire (NCCN distress thermometer) to describe the profiles of the patients in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided